CLINICAL TRIAL: NCT06641232
Title: Comparison of Anesthetic Efficacy and Safety Between Nerve Block and Infiltrative Technique for Mandibular Posterior Implant Placement. a Triple-blind Randomized Clinical Trial.
Brief Title: Comparison of Anesthetic Efficacy and Safety Between Nerve Block and Infiltrative Technique for Mandibular Posterior Implant Placement.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Adrià Jorba García, Prof. dr (DDS, MS,PhD), University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-2024
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-10

CONDITIONS: Dental Implants; Local Anesthesia
Keywords: dental implants; local anesthesia; block nerve

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inferior dental nerve block (Experimental): One articaine cartridge (1.8 mL of articaine 4% at 1:100,000) with the direct technique for the inferior dental nerve block and half a cartridge (0.9 mL) for the buccal nerve block.
  Interventions: Procedure: Comparison of anesthetic efficacy and safety between nerve block and infiltrative technique for mandibular posterior implant placement.
- Infiltrative (Active Comparator): One anesthetic cartridge (1.8 mL of articaine 4% 1:100,000) using the vestibular infiltrative technique (supraperiosteal paraapical). Subsequently administer half a cartridge of anesthetic (0.9 mL of articaine 4% 1:100,000) using the infiltrative technique (supraperiosteal paraapical) lingually in the sublingual area of the tooth to be treated.
  Interventions: Procedure: Comparison of anesthetic efficacy and safety between nerve block and infiltrative technique for mandibular posterior implant placement.

INTERVENTIONS:
Procedure: Comparison of anesthetic efficacy and safety between nerve block and infiltrative technique for mandibular posterior implant placement. — The surgeon and his assistant will leave the operating room and the study investigator in charge of anesthetizing the patients (XA) will enter.
  The anesthesia will be performed by an investigator other than the surgeon performing the procedure. The patient will be assigned to a treatment group; patients in the control group will undergo vestibular and lingual infiltration, while the experimental group will undergo inferior dental nerve block together with buccal nerve block.

SUMMARY:
The goal of this triple blind randomized clinical trial is to compare the safety, efficacy and postoperative pain between the inferior dental nerve block (IDNB) and the infiltrative technique (TINF) in the placement of mandibular posterior dental implants in patients with partial edentulism.

The main questions it aims to answer are:

* The anesthetic efficacy of the IDNB technique, measured as the number of reanesthesias during the surgical procedure, is superior to the infiltrative technique in the placement of dental implants in the posterior mandibular area.
* The IDNB technique presents a higher rate of adverse effects than TINF in the placement of dental implants in the posterior mandibular area.
* The IDNB technique presents less postoperative pain than TINF in the placement of dental implants in the posterior mandibular area.

The investigator (XA) will perform the anesthetic technique. A modified dental anxiety questionnaire (MDAS) will be administered prior to surgery. Then, 2g of Amoxicillin will be administered 1 hour before the surgery. Subsequently, the surgeon and his assistant will prepare the surgical field with sterile sizes. The surgeon and assistant will then leave the operating room and the study investigator in charge of anesthetizing the patients (XA) will enter.

The anesthesia will be performed by an investigator other than the surgeon performing the procedure. The patient will be assigned to a treatment group; patients in the control group will undergo vestibular and lingual infiltration, while the experimental group will undergo IDNB together with buccal nerve block.

The anesthetic latency time will be determined by using a pulpometer on the most posterior tooth in the arch.

Failure to achieve sufficient anesthetic depth, as measured by pulpometer, within 6 minutes of the last puncture will be considered early anesthetic failure and will be counted as such.

* Subsequently, a student of the Master's Degree in Oral Surgery of the University of Barcelona will perform the surgical intervention. The surgeons in charge of performing the surgery will not know to which group each patient belongs.
* The collection of the variables and the postoperative controls will be carried out by the researcher who has not performed the anesthetic technique and who will not know the study group to which the patient belongs.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age (≥18 years), partially edentulous, requiring the placement of one or more mandibular implants in the molar area.
* Patients without relevant systemic pathology (equal or lower than ASA II).
* Sufficient intellectual capacity to understand the study, the informed consent and to adequately complete the questionnaires.

Exclusion Criteria:

* - Pregnant patients.
* Patients with allergy or hypersensitivity to articaine or adrenaline.
* Patients with uncontrolled systemic diseases.
* Patients who may recognize the anesthetic technique used (e.g. dentists).
* Drugs or systemic diseases (ASA III or higher) that contraindicate surgical intervention or the use of anesthetics and/or vasoconstrictors.
* Patients with relative or absolute contraindication of conventional analgesic or anti-inflammatory regimen.
* Immediate implants.
* Surgeries requiring bone grafts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy of the inferior dental nerve block and the infiltrative technique in the placement of mandibular posterior dental implants in patients with partial edentulism. | 1 hour
  Determined by: Reporting a negative response to the pulpometer within 6 minutes after injection. Absence of need for reanesthesia during the surgical procedure.

SECONDARY OUTCOMES:
To evaluate the safety of anesthetic techniques used in the placement of dental implants in the posterior mandibular region. | 7 days
  Determined by the appearance or absence of adverse effects, such as : Disorientation, dizziness, blurred vision, nausea, vomiting, tremors, convulsions, vasovagal syncope, paresthesia or trismus.
To analyze the postoperative pain associated with the placement of mandibular implants using an inferior dental nerve block compared to those implanted with infiltrative techniques. | 7 days
  Determined using a visual anlogical scale of 10 cm at the 2, 6, and 12 hours posteriors to the surgery and then everyday until the 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital odontológic de Bellvitge, Universitat de Barcelona, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garcia-Blanco M, Gualtieri AF, Puia SA. A randomized controlled trial comparing nerve block and mandibular infiltration techniques in posterior mandible implant surgeries. J Clin Exp Dent. 2018 Oct 1;10(10):e1003-e1010. doi: 10.4317/jced.54330. eCollection 2018 Oct. PMID 30386507
- [Background] Heller AA, Shankland WE 2nd. Alternative to the inferior alveolar nerve block anesthesia when placing mandibular dental implants posterior to the mental foramen. J Oral Implantol. 2001;27(3):127-33. doi: 10.1563/1548-1336(2001)0272.3.CO;2. PMID 12500871
- [Background] Esteve-Pardo G, De-Larriva E, Salgado A, Bernabeu-Esclapez A, Bardaji JA, Esteve-Colomina L. Is Inferior Alveolar Nerve Block Needed to Perform Implant Surgery in the Posterior Mandible? A Randomized Controlled Trial. J Oral Maxillofac Surg. 2022 Mar;80(3):490-500. doi: 10.1016/j.joms.2021.09.028. Epub 2021 Oct 10. PMID 34762850
- [Background] Escoda CG, Aytés LB. Tratado De Cirugia Bucal. Anim Genet. 2008;39:561-3.
- [Background] Sanchez-Siles M, Torres-Diez LC, Camacho-Alonso F, Salazar-Sanchez N, Ballester Ferrandis JF. High volume local anesthesia as a postoperative factor of pain and swelling in dental implants. Clin Implant Dent Relat Res. 2014 Jun;16(3):429-34. doi: 10.1111/cid.12005. Epub 2012 Sep 21. PMID 22998596
- [Background] Sancho-Puchades M, Vilchez-Perez MA, Valmaseda-Castellon E, Paredes-Garcia J, Berini-Aytes L, Gay-Escoda C. Bupivacaine 0.5% versus articaine 4% for the removal of lower third molars. A crossover randomized controlled trial. Med Oral Patol Oral Cir Bucal. 2012 May 1;17(3):e462-8. doi: 10.4317/medoral.17628. PMID 22143739
- [Background] Gaffen AS, Haas DA. Retrospective review of voluntary reports of nonsurgical paresthesia in dentistry. J Can Dent Assoc. 2009 Oct;75(8):579. PMID 19840499
- [Background] Garisto GA, Gaffen AS, Lawrence HP, Tenenbaum HC, Haas DA. Occurrence of paresthesia after dental local anesthetic administration in the United States. J Am Dent Assoc. 2010 Jul;141(7):836-44. doi: 10.14219/jada.archive.2010.0281. PMID 20592403
- [Background] Haas DA, Lennon D. A 21 year retrospective study of reports of paresthesia following local anesthetic administration. J Can Dent Assoc. 1995 Apr;61(4):319-20, 323-6, 329-30. PMID 7736335
- [Background] Hillerup S, Jensen R. Nerve injury caused by mandibular block analgesia. Int J Oral Maxillofac Surg. 2006 May;35(5):437-43. doi: 10.1016/j.ijom.2005.10.004. Epub 2005 Dec 15. PMID 16343853
- [Background] Renton T, Janjua H, Gallagher JE, Dalgleish M, Yilmaz Z. UK dentists' experience of iatrogenic trigeminal nerve injuries in relation to routine dental procedures: why, when and how often? Br Dent J. 2013 Jun;214(12):633-42. doi: 10.1038/sj.bdj.2013.583. PMID 23787854
- [Background] Kim C, Hwang KG, Park CJ. Local anesthesia for mandibular third molar extraction. J Dent Anesth Pain Med. 2018 Oct;18(5):287-294. doi: 10.17245/jdapm.2018.18.5.287. Epub 2018 Oct 31. PMID 30402548
- [Background] Camps-Font O, Figueiredo R, Sanchez-Torres A, Cle-Ovejero A, Coulthard P, Gay-Escoda C, Valmaseda-Castellon E. Which is the most suitable local anaesthetic when inferior nerve blocks are used for impacted mandibular third molar extraction? A network meta-analysis. Int J Oral Maxillofac Surg. 2020 Nov;49(11):1497-1507. doi: 10.1016/j.ijom.2020.04.016. Epub 2020 May 27. PMID 32473767
- [Background] Santos-Sanz L, Toledano-Serrabona J, Gay-Escoda C. Safety and efficacy of 4% articaine in mandibular third-molar extraction: A systematic review and meta-analysis of randomized clinical trials. J Am Dent Assoc. 2020 Dec;151(12):912-923.e10. doi: 10.1016/j.adaj.2020.08.016. PMID 33228884
- [Background] Bataineh AB, Alwarafi MA. Patient's pain perception during mandibular molar extraction with articaine: a comparison study between infiltration and inferior alveolar nerve block. Clin Oral Investig. 2016 Nov;20(8):2241-2250. doi: 10.1007/s00784-016-1712-8. Epub 2016 Jan 21. PMID 26791025
- [Background] Albrektsson T, Branemark PI, Hansson HA, Lindstrom J. Osseointegrated titanium implants. Requirements for ensuring a long-lasting, direct bone-to-implant anchorage in man. Acta Orthop Scand. 1981;52(2):155-70. doi: 10.3109/17453678108991776. PMID 7246093
- [Background] Fischer K, Stenberg T. Prospective 10-year cohort study based on a randomized controlled trial (RCT) on implant-supported full-arch maxillary prostheses. Part 1: sandblasted and acid-etched implants and mucosal tissue. Clin Implant Dent Relat Res. 2012 Dec;14(6):808-15. doi: 10.1111/j.1708-8208.2011.00389.x. Epub 2011 Oct 18. PMID 22008715
- [Background] Degidi M, Nardi D, Piattelli A. 10-year follow-up of immediately loaded implants with TiUnite porous anodized surface. Clin Implant Dent Relat Res. 2012 Dec;14(6):828-38. doi: 10.1111/j.1708-8208.2012.00446.x. Epub 2012 Feb 29. PMID 22376174
- [Background] Buser D, Janner SF, Wittneben JG, Bragger U, Ramseier CA, Salvi GE. 10-year survival and success rates of 511 titanium implants with a sandblasted and acid-etched surface: a retrospective study in 303 partially edentulous patients. Clin Implant Dent Relat Res. 2012 Dec;14(6):839-51. doi: 10.1111/j.1708-8208.2012.00456.x. PMID 22897683